CLINICAL TRIAL: NCT00838149
Title: Effect of Glutamine Supplementation on the Structure and Function of the Mucosa of Small Intestine in Crohn's Disease: A Randomized Controlled Trial
Brief Title: Effect of Glutamine on Intestinal Permeability in Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Prof. Y K Joshi, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I458
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Glutamine; Whey Proteins; Whey

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glutamine (Active Comparator): Glutamine would be supplemented (0.5gm/Kg ideal body weight) in the form of a water soluble commercial preparation containing 10 gm of pure L- Glutamine in the crystalline form. The patient in this group would be counseled to meet the remaining protein requirement (i.e1g/Kg/wt) by usual diet. This intervention would be made over a period of two months.
  Interventions: Dietary Supplement: Glutamine
- Whey Protein (Placebo Comparator): Whey Protein:
  Whey protein would be supplemented (0.5gm/Kg ideal body weight) in the form of a water soluble whey protein concentrate containing 70 % protein. The patient in this group would be counseled to meet the remaining protein requirement (i.e1g/Kg/wt) by usual diet. This intervention would be made over a period of two months.
  Interventions: Dietary Supplement: Glutamine; Dietary Supplement: Whey protein

INTERVENTIONS:
Dietary Supplement: Glutamine — Glutamine group :
  Glutamine would be supplemented (0.5gm/Kg ideal body weight) in the form of a water soluble commercial preparation containing 10 gm of pure L- Glutamine in the crystalline form. The patient in this group would be counseled to meet the remaining protein requirement (i.e1g/Kg/wt) by usual diet. This intervention would be made over a period of two months.
  Other Names: L-Glutamine
Dietary Supplement: Whey protein — Whey protein group:
  Whey protein would be supplemented (0.5gm/Kg ideal body weight) in the form of a water soluble whey protein concentrate containing 70 % protein. The patient in this group would be counseled to meet the remaining protein requirement (i.e1g/Kg/wt) by usual diet. This intervention would be made over a period of two months.
  Other Names: Whey Protein Concentrate
  Arms: Whey Protein

SUMMARY:
The purpose of this study is to see whether enteral glutamine supplementation improves intestinal permeability and small intestinal morphology in patients with Crohn's disease.

DETAILED DESCRIPTION:
Glutamine is the most abundant amino acid in the body constituting 50% to 60% of total free amino acid pool in muscle and 20% in plasma. Recently it has been reclassified as a conditionally essential amino acid due to body's inability to synthesize sufficient amount under stressful conditions like trauma and sepsis. It is an essential fuel for fibroblasts, lymphocytes and enterocytes. It plays an important role in nitrogen balance and an integral role in glucose regulation and also in acid base homeostasis. It is an essential ingredient for glutathione, an important antioxidant. During the last decade a number of experimental and clinical studies, by using enteral and parenteral glutamine supplements, have shown its beneficial role in conditions like sepsis and infection, elective surgery and accidental injury, catabolic state, fetal and critically ill low birth weight neonates and cancer. A few experimental and clinical studies have also shown its positive role in inflammatory bowel disease, which is attributed to the effect of glutamine on intestinal permeability, growth of enterocytes, enhancement of gut immunity and glutathione synthesis. So far there is hardly any well-planned randomized trial of enteral glutamine supplements in Crohn's disease. Hence this study is planned to evaluate effect of enteral glutamine supplements on structure and function of intestine in patients with Crohn's disease.

Diagnosed cases of Crohn's Disease attending Gastroenterology OPD or admitted in ward at AIIMS will be randomized into two groups, glutamine and whey protein group. The parameters for intestinal function and structure tested will be, permeability, villous height, plasma glutamine and D-xylose absorption at the base line and at the end of the intervention. As per the available data improvement is expected in both structure and function of the intestine, which will be an important contribution in the management of this chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* All the consecutive patients with Crohn's disease in the remission phase with an abnormal intestinal permeability (IP)

Exclusion Criteria:

* Patients in the active phase of the disease i.e. CDAI score >150
* Patients with a normal intestinal permeability i.e. LMR < 0.0373
* Patients already taking a high protein nutritional supplement
* Patients with other associated systemic diseases like chronic liver disease, chronic kidney disease, diabetes mellitus, malignancy
* Patients with a special physiologic condition i.e., pregnancy or lactation.
* Patients lesser than 15 years (pediatric group) and more than 60 years of age (elderly patients)

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2005-11; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Improvement in intestinal permeability after glutamine supplementation | Baseline and after two months of intervention

SECONDARY OUTCOMES:
Change in small intestinal morphology after glutamine supplementation | Baseline and after two months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yogendra K Joshi, M.D., PhD., Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, New Delhi, India